CLINICAL TRIAL: NCT00780156
Title: The ITALIC Study Is There A LIfe for DES After Discontinuation of Clopidogrel : The ITALIC Study
Brief Title: The ITALIC Study: Is There A LIfe for Drug-eluting Stents (DES) After Discontinuation of Clopidogrel
Acronym: ITALIC
Status: Terminated | Type: Observational
Why Stopped: No more information will be given. No consequences on security and treatment of patients: standard therapy is already performed for all patients.
Sponsor: French Cardiology Society (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 2008-004131-38; 2008-02
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Restenosis
Keywords: Drug eluting stent; Dual antiplatelet therapy; bleeding; stent thrombosis; follow-up of the drug eluting stent
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background

Drug-eluting stents (DES) have been extremely successful in reducing restenosis and the need for repeat revascularization procedures in patients who undergo PCI. The potential increased incidence of late stent thrombosis prompted cardiologists to prolong the use of dual anti-platelet therapy after the one year duration recommended by the recent ESC guidelines. However, while the premise that the cardiologists should put all their patients on dual clopidogrel-aspirin regimen for life sounds the easy way, it is an unrealistic goal because of the potential increase of bleeding complications and of the healthcare cost increase. The recent possibility to monitor aspirin with bedside assays offers a real opportunity to compare in good aspirin responder patients the two strategies: aspirin-clopidogrel regimen versus mono-aspirin regimen and to respond to the key question: can the investigators switch from dual to single antiplatelet therapy after six months in good aspirin responder patients ? Study National, multicenter, randomised prospective open group comparison of dual clopidogrel-ASA versus single ASA regimen after six months, in good ASA responder patients treated with DES (name: XIENCE) implantation.

End point Primary: At 12 months: death, myocardial infarction, repeat urgent revascularization, stroke requiring a new hospitalisation and major bleedings.

Secondary: Incidence at 24 and 36 months after drug eluting stent(name: XIENCE) implantation, of the same composite endpoint and incidence at 12, 24 and 36 months of minor bleeding complications Participating centres: 60 french centers

Date of study beginning: November 2008 Duration of inclusion: 9 months Duration of study: 45 months

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject ≥ 18 years of age eligible for PCI with at least one drug eluting stent (name: Xience) implanted in all clinical situations excluding primary PCI for acute MI and treatment of the left main artery.
* Male or female subject ≥ 18 years of age eligible for PCI with at least one DES Xience.
* Patient not pre-treated with protein IIb/IIIa inhibitors (name: abxicimab or eptifibatide) during hospitalization
* Patient pre-treated with aspirin and clopidogrel before PCI
* ASA check at least 24 hours after the interruption of tirofiban
* The subject has given written informed and dated consent to participate in this study.

Exclusion Criteria:

* Subjects not able to give informed consent
* Prior implantation of DES
* Known platelets < 100 000/µl or known hemorrhagic diathesis
* Oral anticoagulation or treatment with abxicimab or eptifibatide during hospitalization
* ASA check less than 24 hours after the interruption of tirofiban
* Thrombolytic therapy within 4 days before ASA check
* Contra-indication to aspirin or clopidogrel
* Recent major surgery < 6 weeks
* Evidence of an active gastrointestinal or urogenital bleeding
* Severe liver insufficiency
* Primary PCI for acute MI
* Left main PCI
* Any scheduled surgery during the year after enrollment
* Severe concomitant disease with life expectation < two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after drug eluting stent implantation
Sampling Method: Probability Sample
Enrollment: 1235 (Actual)
Dates: Start 2008-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Incidence after XIENCE implantation of a composite endpoint of death, MI, repeat urgent revascularization, stroke requiring a new hospitalisation | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- department Cardiology, Brest, France